CLINICAL TRIAL: NCT03432091
Title: Effects of a Melatonin Receptor Agonist on Clinical Manifestations and Peripheral Biological Markers of Circadian Rhythm
Brief Title: Melatonin Receptor Agonist and Peripheral Biological Markers
Status: Completed | Type: Observational
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuan-Pin, Chief of psychiatry, National Science and Technology Council, Taiwan
Other Study IDs: CMUH104-REC1-105
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Insomnia
Keywords: melatonin; melatonin receptor agonist; circadian-clock-related genes
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The higher values of circadian-clock-related proteins observed at day (brain and muscle aryl hydrocarbon receptor nuclear translocator-like protein 1 and circadian locomoter output cycles protein kaput1) and night (period circadian protein homolog 1 and cryptochrome). Melatonin receptor type 1 (MT1) and melatonin receptor type 2 (MT2) are present in mammals including humans and involved in sleep-wake cycle.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: melatonin — Ramelteon RMT (RMT, Rozerem®), a novel MT1 and MT2 agonist, has been approved for treatment of insomnia, and provides a strong phase shift signal to the circadian timing system. Melatonin receptor agonists have recently become available for treatment of sleep and psychiatric disorders

SUMMARY:
People who have insomnia typically co-occur with mental disorders, especially anxiety and depression. It has been documented that the melatonin phase in the depressed patients was reached with a delay. Melatonin plays a crucial role in regulation of circadian-clock-related gene expression.

DETAILED DESCRIPTION:
The higher values of circadian-clock-related proteins observed at day (brain and muscle aryl hydrocarbon receptor nuclear translocator-like protein 1 and circadian locomoter output cycles protein kaput1) and night (period circadian protein homolog 1 and cryptochrome). Melatonin receptor type 1 (MT1) and melatonin receptor type 2 (MT2) are present in mammals including humans and involved in sleep-wake cycle. RamelteonRMT (RMT, Rozerem®), a novel MT1 and MT2 agonist, has been approved for treatment of insomnia, and provides a strong phase shift signal to the circadian timing system. Melatonin receptor agonists have recently become available for treatment of sleep and psychiatric disorders; however, the effects of the melatonin receptor agonist on peripheral biological markers of circadian rhythm are still to elucidate. This is a non-randomized, observational study, which aims of this study is to evaluate the effects of ramelteon RMT in melatonin level and the regulation of circadian rhythm genes expression in patients with primary insomnia, and/or major depressive disorder (MDD) on, or generalized anxiety disorder (GAD) with symptoms of insomnia. Forty Participants: Participants aged 20-80 years with body mass index between 18 and 34 and without any ambulatory problems will be recruited according to clinical judgment to take RMT for insomnia, ages 20-80 years, body mass index between 18 and 34, without any ambulatory problems, and be willing to write sleep diary. Primary insomnia, MDD and GAD will be as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised for at least 3 months and a history of daytime complaint(s) associated with disturbed sleep. Participants were administered the ramelteon RMT tablet (8 mg/Tab) by oral intake at the same time, which is 2 hours prior to the schedule bedtime every night for eight weeks. The peripheral blood is collected at two time points - ramelteon RMT administration week 0 and week 8, and the melatonin, circadian-clock-related day genes (Aryl hydrocarbon receptor nuclear translocator-like protein 1 and Circadian locomoter output cycles protein kaput1) and night genes (circadian protein homolog 1 and cryptochrome) expression variation will be quantified and compared to determine circadian rhythm phase shift. The expected findings are the circadian-clock-related genes would shift to normal baseline and these genes expressions will be the peripheral marker for evaluation of drug treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Out-patients with primary insomnia and patients with major depressive disorder (MDD) and generalized anxiety disorder (GAD) with chief complaint of insomnia or a history of daytime complaint(s) associated with disturbed sleep. The diagnosis of MDD and GAD will be made made according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) Revised for at least 3 months.
2. Patients are 20-80 years old, body mass index between 18 and 34, and without any ambulatory problems.
3. Subject is a male or a post-menopausal female. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
4. If they willing to give written informed consent and cooperative in this study. They are willing to write sleep diary.
5. Subjective sleep latency greater than or equal to 45 minutes and a subjective total sleep time less than or equal to 6.5 hours per night for at least 3 nights during the week of the lead-in period.
6. Habitual bedtime is between 8:30 PM and 12:00 AM.

Exclusion Criteria:

1. Known hypersensitivity to ramelteon or related compounds, including melatonin.
2. Previously participated in a study involving ramelteon.
3. Participated in any other investigational study, and/or took any investigational drug within 30 days or five half-lives prior to the first day of single-blind study medication, whichever is longer.
4. Sleep schedule changes required by employment (eg, shift worker) within three months prior to the first day of single-blind study medication, or has flown across greater than three time zones within seven days prior to screening.
5. Participated in a weight loss program or substantially altered exercise routine within 30 days prior to the first day of single blind study medication.
6. Has ever had a history of seizures, sleep apnea, chronic obstructive pulmonary disease, restless leg syndrome, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
7. History of substance use disorders, such drug addiction, drug abuse, alcohol abuse within the past 12 months, as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised and/or regularly consumes 4 or more alcoholic drinks per day.
8. History of drug addiction or drug abuse within the past 12 months.
9. Positive hepatitis panels.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Out-patients with primary insomnia and patients with major depressive disorder (MDD) and generalized anxiety disorder (GAD) with chief complaint of insomnia or a history of daytime complaint(s) associated with disturbed sleep. The diagnosis of MDD and GAD will be made made according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) Revised for at least 3 months.
  2. Patients are 20-80 years old, body mass index between 18 and 34, and without any ambulatory problems.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The Change from Baseline Hamilton depression rating scale at 8 weeks | 8 weeks
  This scale scores 0-64 points;The higher total score indicates a more severe

SECONDARY OUTCOMES:
The Change from Baseline pittsburgh sleep quality index rating scale at 8 weeks | 8 weeks
  This scale scores 0-21 points;The higher total score indicates a more severe

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Pin Su, MD PhD, Principal Investigator — China Medical University Hospital

IPD SHARING:
Plan to Share IPD: No